CLINICAL TRIAL: NCT07197021
Title: Transcatheter Edge-to-Edge Repair In Moderate and Exertional-Induced Severe MR (TIMER)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, The first affiliated hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIMER
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Mitral Regurgitation Functional
Keywords: hand grip; TEER; moderate
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEER (Experimental): TEER
  Interventions: Device: TEER; Drug: GDMT
- Control group (Placebo Comparator): GDMT
  Interventions: Drug: GDMT

INTERVENTIONS:
Device: TEER — TEER
  Arms: TEER
Drug: GDMT — GDMT

SUMMARY:
Transcatheter Edge-to-Edge Repair (TEER) has become an established alternative for the treatment of severe mitral regurgitation (MR). RESHAPE trial indicated that patients with moderate functional MR (FMR) and heart failure (HF) might benefit from TEER. However, it still not clear that TEER is effective for which subset of patients with FMR.

Hand-Gripping (HG), characterized with an increased venous return, preservation or increase of left ventricular (LV) afterload and systemic vascular resistance, has been identified as a means of stress test to identify exertion-induced mitral regurgitation. Most importantly, compared to exercise stress testing via treadmill running or cycling in patients with moderate FMR, HG demonstrates significantly higher feasibility and safety.

HG-induced severe MR reflects the reversibility of the regurgitation under stress, suggesting that reducing MR through TEER might alleviate LV volume overload, improve cardiac efficiency, and mitigate symptoms, which need to be validated in this trial.

TIMER is a multi-center, randomized, double blind, placebo-controlled trial. A total of 300 patients with moderate and exertional-induced severe MR will be randomized in a 1:1 ratio to the treatment with TEER and guideline-directed medical therapy (GDMT) or GDMT only.

The primary endpoint of this study is rehospitalization within 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate functional mitral regurgitation
2. HG-induced severe functional mitral regurgitation
3. Left ventricular ejection fraction (LVEF) between 20% to 50%
4. Left ventricular end-systolic diameter (LVESD) ≤70 mm

Exclusion Criteria:

1. Stage D heart failure per ACC/AHA guidelines with hemodynamic instability or cardiogenic shock
2. Untreated symptomatic coronary artery disease requiring revascularization
3. Chronic obstructive pulmonary disease (COPD) requiring continuous oxygen therapy or long-term corticosteroids therapy
4. Severe pulmonary hypertension or moderate-to-severe right ventricular dysfunction
5. Aortic or tricuspid valve disease requiring surgical or transcatheter intervention
6. Life expectancy <12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization rate | 24 months
  Rehospitalization rate within 24 months

SECONDARY OUTCOMES:
KCCQ | 24 months
  Range of 0-100, with higher scores indicating better health status
NYHA class | 24 months
  I-IV
6-min walk test | 24 months
  >500 m: Normal exercise capacity 350-500 m: Mild impairment 150-350 m: Moderate impairment <150 m: Severe impairment
MACE | 24 months
  Cardiovascular Death, Myocardial Infarction, Stroke

OTHER OUTCOMES:
Safety Outcome | 24 months
  Complications of TEER

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giustino G, Camaj A, Kapadia SR, Kar S, Abraham WT, Lindenfeld J, Lim DS, Grayburn PA, Cohen DJ, Redfors B, Zhou Z, Pocock SJ, Asch FM, Mack MJ, Stone GW. Hospitalizations and Mortality in Patients With Secondary Mitral Regurgitation and Heart Failure: The COAPT Trial. J Am Coll Cardiol. 2022 Nov 15;80(20):1857-1868. doi: 10.1016/j.jacc.2022.08.803. PMID 36357085
- [Background] Alachkar MN, Kirschfink A, Grebe J, Almalla M, Frick M, Milzi A, Moersen W, Becker M, Marx N, Altiok E. Dynamic handgrip exercise for the evaluation of mitral valve regurgitation: an echocardiographic study to identify exertion induced severe mitral regurgitation. Int J Cardiovasc Imaging. 2021 Mar;37(3):891-902. doi: 10.1007/s10554-020-02063-5. Epub 2020 Oct 16. PMID 33064244